CLINICAL TRIAL: NCT05479409
Title: Effect of Neoadjuvant Radiation and Prediction of Response to Treatment in Locally Advanced Breast Cancer
Brief Title: Neoadjuvant Radiation in Locally Advanced Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaoli Yu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FDRT-BC016
Record Dates: First submitted 2022-06-29; First posted 2022-07-29 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Breast Neoplasms
Keywords: breast cancer; neoadjuvant radiotherapy; biomarkers
MeSH Terms: conditions — Breast Neoplasms | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Intervention Model Description: Preoperative radiotherapy and concurrent chemotherapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant radiotherapy (Experimental): Group 1:Patients undergo mastectomy or Breast conserving surgery after radiotherapy Group 2:Patients receive boost in the area of residual breast mass and regional lymph node. A total dose of 66Gy will be given.
  Interventions: Radiation: Neoadjuvant radiotherapy

INTERVENTIONS:
Radiation: Neoadjuvant radiotherapy — radiation therapy combined with chemotherapy prior to surgery

SUMMARY:
The purpose of this study is to determine whether neoadjuvant radiation therapy is effective in improving local-regional control and to explore predictors of response to treatment in inoperable breast cancer patients after 2-6 courses of neoadjuvant chemotherapy.

DETAILED DESCRIPTION:
RATIONALE: The optimal management of patients with locally advanced breast cancer(LABC) remains unknown. It is currently accepted that the administration of radiation therapy prior to surgery might result in higher surgery rate or improvement of clinical outcomes.

OUTLINE： This is a prospective phase II study. The purpose is to evaluate the effectiveness of neoadjuvant radiotherapy in combination with chemotherapy. The primary objective in this study is to assess clinical outcomes of these patients. A secondary objective in this study is to identify biomarkers and imaging parameters that can be used as early predictors of treatment response in women with locally advanced breast cancer. Fresh tumor tissue or fresh peripheral blood should be collected as the test sample and stored before treatment. Ultrasound spectroscopy including shear wave elastography parameters should be done before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed locally advanced breast carcinoma
* Inoperable with with 4-6 courses of prior chemotherapy
* No contradiction of radiation or chemo-radiotherapy
* Patients should have the ability to understand and the willingness to sign a written informed consent document
* Signed informed consent must be obtained prior to any study specific procedures

Exclusion Criteria:

* Other prior or concurrent malignancy except adequately treated squamous cell or basal cell skin cancer or contralateral breast DCIS
* Coagulation disorders
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, and cardiac arrhythmia
* Serious underlying medical illness with life expectancy less than 2 years.
* Any condition that is unstable or could jeopardize the safety of the patient and their compliance in the study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Pathological response rate | 1 year
  only for operable patients
Fbjective response rate(ORR) | 3 year
  for inoperable patients
Event free survival(EFS) | 3 year
  for all patients

SECONDARY OUTCOMES:
Time to progression | 3 year
  including local-regional recurrence, disease-free survival, overall survival
Radiation Toxicity | 6 months
  using CTCAE 4.0 and RTOG classification

OTHER OUTCOMES:
Biologic predictor for treatment response | before treatment
  biopsies of the original tumor before treatment for future molecular biology studies in LABC
The role of ultrasound in predicting treatment response | before and 1 month after treatment
  shear wave elastography(SWE) technology

CONTACTS AND LOCATIONS:
Overall Officials: Xiaoli Yu, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No